CLINICAL TRIAL: NCT05939817
Title: The Effect of Intralesian Injection of Umbilical Cord Mesenchymal Stem Cells, Its Conditioned Medium, and Triamcinolone Acetonide on Type 1:3 Collagen Ratio and Interleukin-10 Levels in Keloid: A Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rumah Sakit Pusat Angkatan Darat Gatot Soebroto (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-1206/UN2.F1
Record Dates: First submitted 2023-07-01; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Keloid; Stem Cell
Keywords: Keloid therapy; mesenchymal stem cells; Interleukin-10; collagen ratio
MeSH Terms: conditions — Keloid | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Patients were screened initially by measuring the length and thickness of the keloids using a ruler. Patients who met the study inclusion criteria were randomly divided into 3 groups. Each patient in the groups was given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure. Group 1 was given UC-MSC 2 million cells/mL/cm3, group 2 was given UC-CM 1 mL/cm3, and group 3 was given TA 40 mg/mL/cm3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This double blind, randomized controlled trial (RCT) is carried out according to CONSORT statement. Identical syringes containing the substances were prepared by laboratory staff, in which the researchers were not informed of the syringe contents, in accordance to computerized block randomization. Data processing was then carried out by other statisticians and clinicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- umbilical cord-derived mesenchymal stem cells (UC-MSC) (Experimental): UC-MSC was collected in 50 mL of transport medium, which contained alpha minimal essential medium (αMEM [GIBCO 12000-0221]), penicillin/streptomycin (final concentration 300u/mL [GIBCO 15140-122]) and amphotericin B (final concentration 7500ng /mL [JR Scientific 50701]), and processed in less than 8 hours after collection.
  Group 1 was given UC-MSC 2 million cells/mL/cm3
  Interventions: Biological: umbilical cord-derived mesenchymal stem cells (UC-MSC)
- umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM) (Experimental): group 2 was given UC-CM 1 mL/cm3
  Interventions: Biological: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM)
- triamcinolone acetonide (Active Comparator): group 3 was given TA 40 mg/mL/cm3
  Interventions: Drug: Triamcinolone Acetonide (TA)

INTERVENTIONS:
Biological: umbilical cord-derived mesenchymal stem cells (UC-MSC) — Group 1 was injected UC-MSC 2 million cells/mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: umbilical cord-derived mesenchymal stem cells (UC-MSC)
Biological: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM) — Group 2 was injected UC-CM 1 mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: umbilical cord-derived mesenchymal stem cells conditioned medium (UC-CM)
Drug: Triamcinolone Acetonide (TA) — Group 3 was injected TA 40 mg/mL/cm3, given the same injection volume (1 mL) in every cm3 keloid volume using a 1 mL syringe and 27G needle. The injections were ultrasound-guided into the center of the lesion with a 30-45-degree angle using an in-plane technique, therefore the same pressure.
  Arms: triamcinolone acetonide

SUMMARY:
The objective of this study is to observe the potency of umbilical cord-derived mesenchymal stem cells (UC-MSC) and umbilical cord-derived conditioned medium (UC-CM), or triamcinolone acetonide (TA) in keloid therapy, measured by the decrease in the type 1:3 collagen ratio and the increase of IL-10 levels carried out using CONSORT statement.

DETAILED DESCRIPTION:
Screening of patients were done by measuring keloid dimensions using a ruler. Patients meeting the inclusion criteria were then randomly divided into 3 groups. The same injection volume (1 ml) in every cm3 keloid volume was given using a 1 mL syringe and 27G needle to the subjects. Ultrasound guidance was used to administer the injection using an in-plane technique into the center of the lesion, with inclinations of 30-45 degrees, ensuring uniform pressure in every subject. Group 1 was given UC-MSC 2 million cells/mL/cm3, group 2 receives UC-CM 1mL/cm3 while group 3 was administered TA 40 mg/mL/cm3. In order to obtain UC-MSC and UC-CM, 10 cm of umbilical cord tissue was collected in 50 mL transport medium containing the following substances: amphotericin B (Final concentration 7500 ng/ml [JR Scientific 50701]), alpha minimal essential medium (MEM [GIBCO 12000-022 1]), penicillin/streptomycin (final concentration 300 U/ml [Gibco 15140-122]). Samples were then processed within 8 hours of collection. The umbilical cord was then dissected, briefly washed in 0.5% povidone-iodine (betadine ©) with phosphate buffered saline of pH 7.4 (PBS [Sigma P3813]), and then washed in PBS to remove betadine and blood. The umbilical vessels were excised before the umbilical cord was minced into a complete medium. UC-CM was created using Alpha-MEM and Dulbecco's modified Eagles medium (DMEM [GIBCO 31600-034]). The finalized complete medium contains 1% L-glutamine (Lonza 17-605C), 10% TC (Indonesian Red Cross), amphotericin B (final concentration 2500 ng/ml), and penicillin/streptomycin (final concentration 100 U/ml). Supplementation of culture with 10% autologous or allogeneic cord blood serum and 10% human AB serum (Gibco 34005-100) was done to create MEM. Each well of a 12-well plate (growth are 3.8 cm2 [Biolite]) was filled with three explants (diameter 2-5 mm) and Wharton's Jelly, followed by addition of several drops of complete medium. Triplication of culture was done to each medium. The plate was incubated at 37°C and 5% CO2 and observed daily for contamination or cellular growth, in which the contaminated wells were removed. After the explants was attached, addition of 200-500 µL of appropriate medium was done. Medium changes, involving removal of half of the medium and addition of half of each medium, were performed every 2-3 days. Growth of the cells beyond the explants with 90% confluence marks viability for harvesting using TrypLE Select (GIBCO 12563-011). Dye exclusion method was used to count the viable/non-viable cell yield. After each harvest, with the explant still attached to the plate, new appropriate medium was added with the plate being re-incubated at 37°C and 5% CO2. Similar treatment was repeated for the second and subsequent cultures, enabling multiple harvests from a single explant. Biopsies of the keloid tissues were then conducted twice, in the first meeting and 17 weeks after. Parameters to be evaluated in anatomic pathology examination are Sirius red staining to evaluate collagen structure under a polarizing lens, as well as In Vitro quantitative examination using the ELISA method to examine IL-10. Calculation of changes in the ratio of type 1 to type 3 collagen levels was carried out by dividing the ratio of collagen before treatment from the ratio of collagen after each treatment. When visualized under a polarizing lens, type-3 collagen will appear green-birefringence and type-1 collagen will appear yellow-birefringence. The collagen ratio was obtained by dividing the composition of collagen type 1 to collagen type 3 in Sirius red staining under polarizing lenses.

ELIGIBILITY:
Inclusion Criteria:

* The patient has keloids with a length of 2-10 cm and a thickness of 3-5 mm located on the chest, back, abdomen and extremities
* Patients aged 18 - 55 years
* Post-surgery patients more than 3 months that cause keloids
* The patient is willing to fill in the informed consent form

Exclusion Criteria:

* Patients with hypertrophic scars
* History of kidney failure
* Hypertension
* Pregnant and breastfeeding
* History of blood disorders
* History of tumor or malignancy
* Get other keloid therapy outside of the research procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Type 1:3 collagen ratio reduction | 17 weeks
  Biopsies of the keloid tissues were then conducted twice, in the first meeting and 17 weeks after. Parameters to be evaluated in anatomic pathology examination are Sirius red staining to evaluate collagen structure under a polarizing lens. Calculation of changes in the ratio of type 1 to type 3 collagen levels was carried out by dividing the ratio of collagen before treatment from the ratio of collagen after each treatment. When visualized under a polarizing lens, type-3 collagen will appear green-birefringence and type-1 collagen will appear yellow-birefringence. The collagen ratio was obtained by dividing the composition of collagen type 1 to collagen type 3 in Sirius red staining under polarizing lenses.
IL-10 levels increase | 17 weeks
  Biopsies of the keloid tissues were then conducted twice, in the first meeting and 17 weeks after. Parameters to be evaluated in anatomic pathology examination is In Vitro quantitative examination using the ELISA method to examine IL-10.

CONTACTS AND LOCATIONS:
Locations (1):
- RSPAD Gatot Soebroto, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No